Official Title of the Study

## Clinical Registry Assessment of the Missouri Osteochondral Allograft Preservation System - MOPS

**NCT Number** 

## NCT02503228

Statistical Analysis Plan Updated August 23, 2019

Data were included for statistical analyses when applicable registry data were available for patients undergoing osteochondral and/or meniscal transplantation for the first time (primary transplant) with at least 1-year follow-up data in the registry. Descriptive statistics were calculated to report means, ranges, and percentages. On the basis of the difference in graft preservation methodology, cases were also analyzed by cohort as defined by SP versus MOPS. Chi-square or Fisher exact tests were used to assess for significant differences in proportions. When significant differences in proportions were noted, odds ratios were calculated for relevant comparisons. One-way analysis of variance or t tests were used to assess for significant differences among cohorts at respective time points. Repeated measures analyses of variance were used to assess for significant differences within cohorts over time. Kaplan-Meier survival probability estimates with 95% CIs were calculated and compared. Significance was set at P<.05.